CLINICAL TRIAL: NCT00145509
Title: A Phase 3, Placebo-Controlled, Double-Blinded Continuation Trial Evaluating the Safety and Efficacy of Asenapine in Subjects Completing a 12-week Lead-in Trial and Continuing Lithium or Valproic Acid/Divalproex Sodium for the Treatment of an Acute Manic or Mixed Episode
Brief Title: 40 Week Trial to Study the Safety of Asenapine When Added to Lithium or Valproate in the Treatment of Bipolar Disorder (A7501009)(P05786)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05786; A7501009
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2010-04-16 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asenapine (Active Comparator): Asenapine
  Interventions: Drug: Asenapine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asenapine — Asenapine 5 or 10 mg twice daily (BID) sublingually for 40 weeks
  Other Names: Org 5222
  Arms: Asenapine
Drug: Placebo — Fast-dissolving tablet; twice daily (BID) sublingually for 40 weeks
  Arms: Placebo

SUMMARY:
The primary objective of this trial was to characterize the long-term (up to 40 weeks) safety and tolerability of asenapine in bipolar I disorder subjects who had not completely responded to continuing treatment with lithium or valproic acid (VPA) for the treatment of an acute manic or mixed episodes upon enrollment into the 12-week lead-in trial, A7501008 (NCT00145470). The safety comparison was between the group receiving lithium or VPA and placebo against the group receiving lithium or VPA and asenapine, with the caveat that all subjects may have received benzodiazepine and/or antidepressant rescue medication as needed.

ELIGIBILITY:
Inclusion Criteria:

* Have bipolar I disorder (current episode manic or mixed), be treated with lithium or valproic acid, and have completed the a 12-week lead-in trial

Exclusion Criteria:

* Have an unstable medical condition or clinically significant laboratory abnormality.
* Have a primary diagnosis other than bipolar I disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

REFERENCES:
- [Result] Szegedi A, Calabrese JR, Stet L, Mackle M, Zhao J, Panagides J; Apollo Study Group. Asenapine as adjunctive treatment for acute mania associated with bipolar disorder: results of a 12-week core study and 40-week extension. J Clin Psychopharmacol. 2012 Feb;32(1):46-55. doi: 10.1097/JCP.0b013e31823f872f. PMID 22198448

RESULTS

PARTICIPANT FLOW:
Groups:
- Asenapine: Asenapine 5 or 10 mg sublingually twice daily (BID)
- Placebo: Placebo sublingually BID
Period: Overall Study
Arm/Group | Asenapine | Placebo
Started | 41 | 36
Completed | 19 | 15
Not Completed | 22 | 21
Not completed — Adverse Event | 10 | 3
Not completed — Lack of Efficacy | 3 | 1
Not completed — Lost to Follow-up | 5 | 9
Not completed — Withdrew Consent | 2 | 7
Not completed — Reason not provided | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asenapine | Placebo | Total
Number analyzed (Participants) | 41 | 36 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (11.79) | 38.7 (13.42) | 38.9 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 25 | 18 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: Participants who experienced treatment-emergent adverse events, defined as adverse events reported on or after the first dose of study medication in the 12-week lead-in study through the last dose of study drug + 7 days (or + 30 days for serious adverse events).
Time Frame: up to 52 weeks
Measure: Number; unit: Participants
Arm/Group | Asenapine | Placebo
Number analyzed (Participants) | 41 | 36
Participants | 32 | 25

2. Primary Outcome: Number of Participants Who Discontinued Because of an Adverse Event
Description: Participants who discontinued study medication due to adverse events.
Time Frame: 40 weeks
Measure: Number; unit: participants
Arm/Group | Asenapine | Placebo
Number analyzed (Participants) | 41 | 36
participants | 10 | 3

3. Primary Outcome: Change From Baseline to Week 52 on the Young-Mania Rating Scale (Y-MRS) Score
Description: The Y-MRS is an 11-item, clinician-rated instrument used for assessing the symptoms of mania. Y-MRS total score range = 0-60; higher scores indicate greater severity of symptoms.
Time Frame: Baseline and 52 Weeks
Population: Intent-to-treat are subjects who took at least one dose of double-blind study medication in the extension study and had at least one Y-MRS and MADRS assessment during the extension study.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Asenapine | Placebo
Number analyzed (Participants) | 38 | 33
Score on a Scale | -17.2 (13.65) | -19.7 (11.81)

4. Primary Outcome: Change From Baseline to Week 52 on the Montgomery Asberg Depression Rating Scale (MADRS) Score
Description: The MADRS is a 10-item clinician-rated scale for assessing the severity of symptoms of depression. MADRS total score range = 0-60; higher scores indicate greater severity of symptoms.
Time Frame: Baseline and 52 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Asenapine | Placebo
Number analyzed (Participants) | 38 | 33
Score on a scale | -3.3 (9.75) | -3.9 (7.71)

ADVERSE EVENTS:
Arm/Group | Asenapine | Placebo
Serious Adverse Events (participants affected / at risk) | 9/41 | 4/36
Other Adverse Events (participants affected / at risk) | 25/41 | 18/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=41) | Placebo (N=36)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
BIPOLAR I DISORDER (Psychiatric disorders) | 0 (0) | 1 (3)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSIVE SYMPTOM (Psychiatric disorders) | 1 (1) | 0 (0)
MANIA (Psychiatric disorders) | 4 (4) | 4 (4)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 2 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=41) | Placebo (N=36)
CONSTIPATION (Gastrointestinal disorders) | 4 (8) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 5 (5)
DRY MOUTH (Gastrointestinal disorders) | 3 (3) | 3 (3)
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 3 (3) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (4) | 2 (2)
VOMITING (Gastrointestinal disorders) | 4 (4) | 2 (3)
IRRITABILITY (General disorders) | 3 (3) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (5) | 2 (2)
DIZZINESS (Nervous system disorders) | 2 (2) | 2 (3)
DYSKINESIA (Nervous system disorders) | 3 (4) | 0 (0)
HEADACHE (Nervous system disorders) | 8 (11) | 6 (7)
PARKINSONISM (Nervous system disorders) | 1 (2) | 2 (3)
SEDATION (Nervous system disorders) | 6 (8) | 2 (2)
SOMNOLENCE (Nervous system disorders) | 6 (7) | 3 (4)
TREMOR (Nervous system disorders) | 3 (5) | 3 (3)
ANXIETY (Psychiatric disorders) | 4 (4) | 4 (11)
DEPRESSION (Psychiatric disorders) | 1 (1) | 2 (3)
INSOMNIA (Psychiatric disorders) | 8 (10) | 5 (8)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution will provide manuscripts, abstracts, or the full text of any other intended disclosure to the sponsor at least 30 days prior to submission for publication or other disclosure. If any patent action is required to protect intellectual property rights, Institution agrees to delay the disclosure for a period not to exceed and additional 60 days. Institution will, on request, remove any previously undisclosed Confidential Information (other than study results) before disclosure.